CLINICAL TRIAL: NCT00004357
Title: Phase II Study of Prednisolone/Methylprednisolone Absorption in Children With Juvenile Dermatomyositis
Brief Title: Absorption of Corticosteroids in Children With Juvenile Dermatomyositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Lauren Pachman MD, Children's Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/11924; NU-465
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Vasculitis, Hypersensitivity; Connective Tissue Diseases; Dermatomyositis; Vasculitis
Keywords: Cardiovascular Disease; Respiratory Disease; Rare Diseases; Vasculitis
MeSH Terms: conditions — Vasculitis, Leukocytoclastic, Cutaneous; Connective Tissue Diseases; Dermatomyositis; Vasculitis; Cardiovascular Diseases; Respiration Disorders; Rare Diseases | interventions — Methylprednisolone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methylprednisolone — IV
Drug: Prednisolone — Oral

SUMMARY:
Juvenile dermatomyositis (JDM) is a connective tissue disease that causes skin rash and weak muscles in children. The purpose of this study is to measure the absorption of oral prednisolone and intravenous (IV) methylprednisolone and to determine levels of disease activity indicators in the blood. These levels will be compared to see if there are patterns specific to active and less active JDM.

DETAILED DESCRIPTION:
JDM is a connective tissue disease that is characterized by inflammation of the muscles and the skin. Corticosteroids, such as prednisolone and methylprednisolone, can be administered to help control symptoms of the disease, but absorption patterns of these medications in oral and IV forms are unknown. This study will assess absorption of oral prednisolone and IV methylprednisolone, measure levels of two disease activity indicators (von Willebrand factor and neopterin), and correlate these values in children with JDM.

Patients will participate in this study twice within a period of up to a year, once when the patient's disease is active, and again 6 to 12 months later when the disease is less active. Each of the two study periods will last two nights and two days. Patients will be admitted to the hospital the first night, and a small IV port will be inserted in the patient's arm the first morning to allow for multiple blood draws without additional needle sticks. Patients will receive oral prednisolone the first morning and IV methylprednisolone the second morning. Baseline blood draws will be performed prior to administration of drug, with 13 additional draws over a 6 hour period following drug administration. Following the final blood draw on the second day, the IV port will be removed from the patient's arm and the patient will be discharged from the hospital.

Blood drawn from patients will be assessed for absorption of the drugs and levels of von Willebrand factor and neopterin. Patients will undergo the same sequence of events sometime between 6 to 12 months after the first hospitalization, after their vasculitis is judged to be less active.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile dermatomyositis with evidence of active vasculitis
* Elevated von Willebrand factor antigen prior to study entry
* Elevated neopterin level prior to study entry

Exclusion Criteria:

* Severe renal involvement
* Critically ill or clinically unstable
* Diseases other than dermatomyositis with vasculitis

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 1997-09; Primary Completion 2005-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Pachman, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Children's Memorial Hospital, Chicago, Chicago, Illinois, United States